CLINICAL TRIAL: NCT03836586
Title: Contribution of Pain Catastrophizing to Race Group Differences in Pain and Pain-Related Brain Responses in Older Adults With Knee Osteoarthritis (OA)
Brief Title: Study of Pain Catastrophizing
Acronym: SPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB201802819 -N; P30AG059297 (NIH); K22NS102334 (NIH)
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2022-11

CONDITIONS: Osteo Arthritis Knee
Keywords: catastrophizing; cognitive-behavior therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a single session cognitive-behavioral intervention to reduce pain catastrophizing or a pain education control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Catastrophizing Reduction Group (Experimental): This group will be assigned to a 30-minute, single-session cognitive-behavioral intervention designed to reduce pain catastrophizing.
  Interventions: Behavioral: Cognitive-Behavioral Intervention
- Pain Education Group (Active Comparator): This group will receive general information about the neurobiology of pain and knee OA.
  Interventions: Behavioral: Pain Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Intervention — This intervention comprises three components: 1) general education about pain (e.g., pain pathways) and a rationale for the intervention (e.g., gate control theory); 2) impact of positive and negative pain-related thoughts on neural process of pain; and 3) a guided imaginal pain exposure exercise.
  Arms: Pain Catastrophizing Reduction Group
Behavioral: Pain Education — General information about the neurobiology of pain and knee osteoarthritis will be given to participants assigned to this intervention.
  Arms: Pain Education Group

SUMMARY:
This study proposes to experimentally manipulate pain catastrophizing in order to investigate the neural mechanisms by which pain catastrophizing influences the experience of pain among non-Hispanic Blacks (NHBs) and non- Hispanic Whites (NHWs) with knee osteoarthritis (OA). Therefore, participants will be randomized to either a single session cognitive-behavioral intervention to reduce pain catastrophizing or a pain education control group.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee OA

Exclusion Criteria:

* Younger than 45 years of age or older than 85 years of age
* Prosthetic knee replacement or other clinically significant surgery to the arthritic knee
* uncontrolled hypertension (>150/95)
* Heart disease including heart failure
* Peripheral neuropathy in which pain testing was contraindicated
* Systemic rheumatic disorders including rheumatoid arthritis, systemic lupus erythematosus, gout, and fibromyalgia
* Neurological diseases such as Parkinson's, multiple sclerosis, stroke with loss of sensory or motor function, or uncontrolled seizures
* Significantly greater pain in body sites other than in the knee
* Daily opioid use
* Hospitalization within the preceding year for psychiatric illness
* Currently pregnant or nursing/breastfeeding

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Terry, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pain Catastrophizing Reduction Group | Pain Education Group
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Catastrophizing Reduction Group | Pain Education Group | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.80 (6.83) | 64.20 (6.14) | 60.50 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-Hispanic Black | 2 | 3 | 5
  non-Hispanic White | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Catastrophizing Scale (PCS) at Day 2
Description: 13-item scale that assesses catastrophic thinking associated with pain. The study team will administer the PCS using traditional instructions (a measure of trait catastrophizing) and instructions to assess situation-specific catastrophizing ("Thinking back to your experience during the laboratory pain testing"). Thoughts and feelings concerning pain are ranked on a 0-4 scale, with 0 being the patient has this thought/feeling 'not at all' to 4, the patient has this thought feeling 'all the time.' The PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0 - 52. Higher scores indicate the presence of catastrophizing and therefore worse outcome.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Catastrophizing Reduction Group | Pain Education Group
Number analyzed (Participants) | 5 | 5
score on a scale | 20.40 (25.38) | 15.25 (16.03)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected an average of 2 weeks.
Description: The cognitive-behavioral intervention posed minimal risk to participants.
Arm/Group | Pain Catastrophizing Reduction Group | Pain Education Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT03836586/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03836586/ICF_001.pdf